CLINICAL TRIAL: NCT06435143
Title: Validation and Usability Study of Intermittent Electrical Simulation (Prelivia) IES in the Management of Pressure Injuries Stage 1 and Stage 2
Brief Title: Validation and Usability Study of Intermittent Electrical Simulation in Management of Pressure Injuries Stages 1 and 2
Acronym: IESPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Lisa Maks, Diabetes Clinical Nurse Specialist, Adjunct Professor UBC School of Nursing, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H24-00304
Record Dates: First submitted 2024-05-09; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: This is a feasibility study of testing Prelivia in an in-patient setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with pressure injury stage 1 and stage 2 (Other): Patient admitted to hospital with a confirmed stage 1 and 2 pressure injuries. Prelivia device will be applied to skin around pressure injury. Intermittent electrical stimulation will be administered for 10 seconds every 10 minutes to improve blood flow and muscle contraction to the area, simulating movement
  Interventions: Device: Prelivia

INTERVENTIONS:
Device: Prelivia — Pad applied to skin provide electrical stimulation for 10 seconds every 10 minutes
  Other Names: Intermittent electrical stimulation

SUMMARY:
The focus of this study will be early stage pressure ulcers, which can quickly progress to stage 3, 4 or deep tissue injury The proposed study explores the feasibility of intermittent electrical stimulation (IES),Prelivia, a novel, non-invasive technology in the management of stage 1 and 2 pressure ulcers.

DETAILED DESCRIPTION:
Pressure ulcers (also known as pressure injuries or bedsores) constitute a major morbidity in critically ill patients due to immobilization, deranged tissue perfusion, and poor nutrition. It is estimated that the prevalence of pressure injuries is 2.2 to 23.9 percent or higher, depending on the hospital environment, significantly contributing to nosocomial risk and healthcare costs.

Particularly, they are one of the most common complications among people with limited mobility is increased pressure on certain areas of the body causing reduced blood flow and damage to the skin.

There has been extensive research that shows electrical stimulation can be useful in pressure ulcer treatment. (Arora et al, 2020) (5) Electrical stimulation is provided by an electrical current, which can be applied in many ways.

The study intervention applies Intermittent Electrical Stimulation (IES) to the affected area through surface electrodes. The device invokes muscle contractions for 10 seconds every 10 minutes, emulating the subconscious adjustments performed by able- bodied individuals in response to discomfort when seated or lying down. Animal studies demonstrate that IES reduces internal pressure at bone-muscle interfaces (the hypothesized mechanism for injury development), increases tissue oxygenation in surrounding areas, and reduces or eliminates deep tissue injury in muscles subjected to prolonged loading (Appendix A). (6) (L. Solis et al., 2008) (7) Clinical studies support the safety, feasibility, and general acceptability of gluteal IES in human participants. (Appendix B) (Ahmetovic et al., 2015) (8) (Kane et al., 2017) (9) This technology has been studied and has shown, with strong evidence, the capacity of IES to prevent sacral and ischial pressure injuries.

Prelivia uses RHT's patented Intermittent Electrical Stimulation (IES) technology which counteracts damaging tissue compression and increases blood flow to parts of the body that are at risk. Prelivia acts by mimicking the physiological micro-contractions that normally occur in mobile individuals when they fidget or shift their weight. Prelivia works by restoring subconscious muscle contractions and movements, or a 'fidgeting' movement that able-bodied individuals are able do. These muscle contractions increase tissue perfusion - the process in which metabolic waste is removed and fresh blood, oxygen, and nutrients are brought into the tissue. The target muscles(such as the glutei maximi) are electrically stimulated for 10 seconds every 10 minutes to restore adequate tissue perfusion to the surrounding tissue.

The system consists of a battery-powered stimulator (Prelivia Stimulator) and disposable hydrogel electrodes. Prelivia's streamlined design, simple application, and low cost make it the ideal addition to existing standard of care procedures.

Prelivia is the only device on the market that addresses poor circulation and low oxygenation in compressed areas. Current pressure injury preventative interventions rely on either temporarily relieving pressure (nurses turn patients every 2 hrs) , creams, or redistributing pressure (specialized mattresses, cushions, etc.). However, neither of these interventions restore blood circulation, tissue oxygenation, or tissue perfusion.

Primary objective: To evaluate users' interaction with the device, safety and tolerability by patients when wearing Prelivia IES during management of pressure injuries stage 1 and 2 during their stay in the hospital, up to 30 days, until patient death or discharge whatever comes first.

Secondary objective : Compare the status and healing time of stage 1 and 2 pressure injuries matched with the historic controls, via retrospective data review. Historic controls will involve consideration of various factors:

Patients with documented stage 1 and 2 pressure injuries matched according to the age range, gender, location of pressure injury(ies), Body mass Index and comorbidities.

Data will be requested from the Providence Healthcare Integrated Health informatics Datalab.

Exploratory objective: Develop high level health economic model for pressure injury cost savings.

ELIGIBILITY:
Inclusion Criteria: Willing and able to provide written informed consent to participate and wear Prelivia for the duration of the study but not longer than 30 days Patients with new or already established stage 1 and 2 pressure injuries BMI <40 Pressure injury location sacral/ischial region

-

Exclusion Criteria:

* existing pressure injury above stage 2 and injuries classified as DTI or unstageable continuous neuromuscular blocking drugs & myasthenia gravis: may prevent the ability of IES to induce muscular contraction
* electrical stimulation to induce muscular contraction
* presence of permanent pacemaker or AICD, and for those with external wires after cardiac surgery, those who are using or at high risk for the development of a requirement for an external pacemaker
* unstable spinal, pelvic, or hop fractures that may be displaced by a forced contraction (for sacral and ischial ulcers)
* rhabdomyolysis
* skin breakdown or malignant skin involvement over the effected regions that would preclude the use of surface electrodes
* any implantable electrostimulation device
* have pacemaker or any other implantable neurostimulation devices,
* if your pressure injury is above stage 2, or
* if you are receiving neuromuscular blocking drugs,
* if you have myasthenia gravis,
* if you have unstable spinal, pelvic, or hip fractures that may be displaced by a forced contraction or
* if you are wearing an incontinence brief and have frequently loose bowel movements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate users' interaction with the device, safety and tolerability by patients when wearing Prelivia IES during management of pressure injuries stage 1 and 2 during their stay in the hospital | 30 days
  Will assess using qualitative questionnaire for both nursing staff and patient as to comfort and ease of use.
Compare the status and healing time of stage 1 and 2 pressure injuries matched with historical controls via retrospective data review. Historic controls will involve consideration of a various factors: | 30 days
  Will perform an initial assessment of the wound (e.g. size, narrative description) and compare this pre-intervention with post-intervention after a maximum of 30 days of wear time.
Exploratory objective: to develop high level health economic model for pressure injury cost savings | 120 days
  Measurement of cost to treat patients that developed a severe pressure ulcer compared to those that did not.

IPD SHARING:
Plan to Share IPD: No
Unidentifyable research data will be shared with other team members